CLINICAL TRIAL: NCT02053363
Title: Low Versus High Dose Tranexamic Acid in Adult Spinal Deformity Surgery: A Randomized, Blinded, Controlled Trial
Brief Title: Tranexamic Acid Dosing in Adult Spinal Deformity Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: AOSpine North America (Industry)
Responsible Party: Principal Investigator, Michael Kelly, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201312010
Record Dates: First submitted 2014-01-28; First posted 2014-02-03 (Estimated); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Adult Spinal Deformity
Keywords: tranexamic acid, reconstructive spine surgery
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Dose/Study Group (Experimental): Tranexamic Acid (Cyklokapron) Loading Dose 50mg/kg given over 15 minutes, followed by 5mg/kg/hr via continuous infusion. The loading dose will be given to coincide with incision. The continuous infusion will be stopped at the conclusion of fascial layer closure.
  Interventions: Drug: Tranexamic Acid (Cyklokapron)
- Standard of Care/Control (Active Comparator): Tranexamic Acid (Cyklokapron) Loading Dose 10mg/kg given over 15 minutes, followed by 1mg/kg/hr via continuous infusion. The loading dose will be given to coincide with incision. The continuous infusion will be stopped at the conclusion of fascial layer closure.
  Interventions: Drug: Tranexamic Acid (Cyklokapron)

INTERVENTIONS:
Drug: Tranexamic Acid (Cyklokapron)

SUMMARY:
The purpose of this study is to evaluate two dosing protocols for tranexamic acid (TXA), an anti-fibrinolytic used to decrease blood loss in adult patients undergoing complex, reconstructive spinal fusion surgeries.

DETAILED DESCRIPTION:
After consent is obtained and the patient is enrolled in the trial, patients will be assigned de-identified, unique identification (ID) numbers. Randomization of these IDs to either low or high dose TXA will occur via a computer generated random assignment. Given the variations that may exist in surgical technique (e.g. performance of osteotomies), stratified randomization will be performed by attending surgeon. Based upon the randomization, the pharmacy will prepare TXA for one of two intravenous dosing protocols:

1. Low Dose (Standard of Care/Control): Loading Dose 10mg/kg given over 15 minutes, followed by 1mg/kg/hr via continuous infusion
2. High Dose (Study Group): Loading Dose 50mg/kg given over 15 minutes, followed by 5mg/kg/hr via continuous infusion.

The surgeon, anesthesia team, and operating room staff will be blind to the concentration of TXA in the medications received. Treatments may be "unblinded" at the discretion of the surgeon and anesthesiologist, in cases of extreme blood loss. If additional anti-fibrinolytics are given, the change in dose will be recorded.

Post-operative care will be the same as any other patient and data collection will be information contained in the patient's medical record that is part of routine, standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (ages 18-75) scheduled to undergo long segment (greater than 8 motion segments) posterior spinal fusion with instrumentation (PSF) for adult scoliosis

Exclusion Criteria:

* Patients with acquired defective color vision
* Subarachnoid hemorrhage
* Active intravascular clotting
* Hypersensitivity to tranexamic acid or any of the ingredients
* Patients who pre-donate autologous blood for intra- or post-operative use (Directed donor units are acceptable)
* History of suspected blood disorders or abnormal coagulation laboratory results
* Current anticoagulation therapy that cannot be interrupted
* History of deep vein thrombosis (DVT)
* Impaired renal function or creatinine clearance <60 ml/min
* Pregnancy or women who are lactating/breastfeeding
* Women on hormonal contraceptives

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Kelly, MD, MSCI(p), Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Baldus CR, Bridwell KH, Lenke LG, Okubadejo GO. Can we safely reduce blood loss during lumbar pedicle subtraction osteotomy procedures using tranexamic acid or aprotinin? A comparative study with controls. Spine (Phila Pa 1976). 2010 Jan 15;35(2):235-9. doi: 10.1097/BRS.0b013e3181c86cb9. PMID 20081519
- [Background] Neilipovitz DT. Tranexamic acid for major spinal surgery. Eur Spine J. 2004 Oct;13 Suppl 1(Suppl 1):S62-5. doi: 10.1007/s00586-004-0716-2. Epub 2004 May 4. PMID 15127250
- [Background] Okubadejo GO, Bridwell KH, Lenke LG, Buchowski JM, Fang DD, Baldus CR, Nielsen CH, Lee CC. Aprotinin may decrease blood loss in complex adult spinal deformity surgery, but it may also increase the risk of acute renal failure. Spine (Phila Pa 1976). 2007 Sep 15;32(20):2265-71. doi: 10.1097/BRS.0b013e31814ce9b0. PMID 17873821
- [Background] Berenholtz SM, Pham JC, Garrett-Mayer E, Atchison CW, Kostuik JP, Cohen DB, Nundy S, Dorman T, Ness PM, Klag MJ, Pronovost PJ, Kebaish KM. Effect of epsilon aminocaproic acid on red-cell transfusion requirements in major spinal surgery. Spine (Phila Pa 1976). 2009 Sep 1;34(19):2096-103. doi: 10.1097/BRS.0b013e3181b1fab2. PMID 19730217
- [Background] Elwatidy S, Jamjoom Z, Elgamal E, Zakaria A, Turkistani A, El-Dawlatly A. Efficacy and safety of prophylactic large dose of tranexamic acid in spine surgery: a prospective, randomized, double-blind, placebo-controlled study. Spine (Phila Pa 1976). 2008 Nov 15;33(24):2577-80. doi: 10.1097/BRS.0b013e318188b9c5. PMID 19011538
- [Background] Gill JB, Chin Y, Levin A, Feng D. The use of antifibrinolytic agents in spine surgery. A meta-analysis. J Bone Joint Surg Am. 2008 Nov;90(11):2399-407. doi: 10.2106/JBJS.G.01179. PMID 18978408
- [Background] Neilipovitz DT, Murto K, Hall L, Barrowman NJ, Splinter WM. A randomized trial of tranexamic acid to reduce blood transfusion for scoliosis surgery. Anesth Analg. 2001 Jul;93(1):82-7. doi: 10.1097/00000539-200107000-00018. PMID 11429344
- [Background] Sethna NF, Zurakowski D, Brustowicz RM, Bacsik J, Sullivan LJ, Shapiro F. Tranexamic acid reduces intraoperative blood loss in pediatric patients undergoing scoliosis surgery. Anesthesiology. 2005 Apr;102(4):727-32. doi: 10.1097/00000542-200504000-00006. PMID 15791100
- [Background] Shapiro F, Zurakowski D, Sethna NF. Tranexamic acid diminishes intraoperative blood loss and transfusion in spinal fusions for duchenne muscular dystrophy scoliosis. Spine (Phila Pa 1976). 2007 Sep 15;32(20):2278-83. doi: 10.1097/BRS.0b013e31814cf139. PMID 17873823
- [Background] Grant JA, Howard J, Luntley J, Harder J, Aleissa S, Parsons D. Perioperative blood transfusion requirements in pediatric scoliosis surgery: the efficacy of tranexamic acid. J Pediatr Orthop. 2009 Apr-May;29(3):300-4. doi: 10.1097/BPO.0b013e31819a85de. PMID 19305284
- [Background] Goobie SM, Meier PM, Pereira LM, McGowan FX, Prescilla RP, Scharp LA, Rogers GF, Proctor MR, Meara JG, Soriano SG, Zurakowski D, Sethna NF. Efficacy of tranexamic acid in pediatric craniosynostosis surgery: a double-blind, placebo-controlled trial. Anesthesiology. 2011 Apr;114(4):862-71. doi: 10.1097/ALN.0b013e318210fd8f. PMID 21364458
- [Derived] Clohisy JCF, Lenke LG, Dafrawy MHE, Wolfe RC, Frazier E, Kelly MP. Randomized, controlled trial of two tranexamic acid dosing protocols in adult spinal deformity surgery. Spine Deform. 2022 Nov;10(6):1399-1406. doi: 10.1007/s43390-022-00539-z. Epub 2022 Jun 25. PMID 35751772

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 Patients consented to participation but withdrew prior to randomization and treatment assignment. Patients either elected not to proceed with the study, did not have surgery, or the proposed surgeries were changed and they were no longer eligible for participation.
Groups:
- High Dose/Study Group: Tranexamic Acid (Cyklokapron) Loading Dose 50mg/kg given over 15 minutes, followed by 5mg/kg/hr via continuous infusion. The loading dose will be given to coincide with incision. The continuous infusion will be stopped at the conclusion of fascial layer closure.
  Tranexamic Acid (Cyklokapron)
- Standard of Care/Control: Tranexamic Acid (Cyklokapron) Loading Dose 10mg/kg given over 15 minutes, followed by 1mg/kg/hr via continuous infusion. The loading dose will be given to coincide with incision. The continuous infusion will be stopped at the conclusion of fascial layer closure.
  Tranexamic Acid (Cyklokapron)
Period: Overall Study
Arm/Group | High Dose/Study Group | Standard of Care/Control
Started | 25 | 27
Completed | 25 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 64 Patients consented to participation. 52 pursued surgery and were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose/Study Group | Standard of Care/Control | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 18 | 34
  >=65 years | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (9.6) | 56.7 (14.3) | 58.3 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 23 | 37
  Male | 11 | 4 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 27 | 52

OUTCOME MEASURES:

1. Primary Outcome: Blood Loss
Description: To compare the estimated blood loss in patients undergoing complex, reconstructive, spinal fusion surgeries receiving one of two dosing protocols for the anti-fibrinolytic, TXA.
  Estimated blood loss was calculated by suction canister volume minus intraoperative irrigation fluid plus blood content in sponges as estimated by weight for all cases.
Time Frame: This outcome is measured during surgery, from exposure to wound closure, approximately 8 hours.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | High Dose/Study Group | Standard of Care/Control
Number analyzed (Participants) | 25 | 27
mL | 2046 (1104) | 1596 (933)

2. Secondary Outcome: Red Blood Cell Transfusions
Description: To compare the mean volume (mL) of packed red blood cell (PRBC) transfusions given to the two groups. Volumes of RBC vary from bag to bag and real volumes will be recorded as provided by the blood bank.
Time Frame: Participants will be followed for the duration of their hospital stay measured from day of surgery to day of discharge from the hospital, approximately 7 days.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | High Dose/Study Group | Standard of Care/Control
Number analyzed (Participants) | 25 | 27
mL | 1259 (868) | 935 (630)

3. Secondary Outcome: Number of Patients Sustaining Intraoperative or 90 Day Complications
Description: To compare the rates of intraoperative complications and 90 day complications observed in the two groups.
Time Frame: Perioperative complications were defined as complications occurring within 90 days of surgery.
Population: All patients achieved 90 day followup
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose/Study Group | Standard of Care/Control
Number analyzed (Participants) | 25 | 27
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: Up to three months after surgery
Arm/Group | High Dose/Study Group | Standard of Care/Control
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 2/25 | 3/27
Other Adverse Events (participants affected / at risk) | 3/25 | 4/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose/Study Group (N=25) | Standard of Care/Control (N=27)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Venothromboembolic Event (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — Deep Vein Thrombosis/Pulmonary Embolism (DVT/PE)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose/Study Group (N=25) | Standard of Care/Control (N=27)
Infection (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Delirium (Nervous system disorders) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Our sample size estimation underestimated the standard deviation of mean EBL in both groups. This resulted in an underpowered study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT02053363/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT02053363/SAP_001.pdf